CLINICAL TRIAL: NCT05823155
Title: Impact of Pre-operative Penicillin Allergy Evaluation on Surgical Prophylaxis: a Randomized Controlled Trial
Brief Title: Impact of Pre-operative Penicillin Allergy Evaluation on Surgical Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Penicillin allergy Protocol V1
Record Dates: First submitted 2022-08-11; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Penicillin Allergy; Surgical Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Detailed penicillin allergy evaluation during pre-operative care (Experimental): This group will undergo a detailed penicillin allergy evaluation performed by an Infectious Diseases specialist. Patients with negative result in skin test and oral provocation test will have their prior labelled penicillin allergy removed from electronic health record, and an additional entry documenting the negative allergy evaluation will be added. A letter signed by an infectious disease specialist documenting the allergy evaluation results will also be given to patients.
  Interventions: Procedure: Detailed penicillin allergy evaluation
- Standard pre-operative care (No Intervention): This group will receive standard perioperative care. The choice of antibiotics during the perioperative period will be decided by surgical team.

INTERVENTIONS:
Procedure: Detailed penicillin allergy evaluation — The intervention group will undergo a detailed penicillin allergy evaluation performed by an Infectious Diseases specialist. Components of penicillin allergy evaluation include verification of allergy history (drug involved including dose and route of administration, exact manifestation of labelled allergy and timing of occurrence after use of alleged culprit, history of skin tests or in vitro testing for diagnosis of allergy, subsequent rechallenge of the same or similar antibiotics), followed by skin test (prick test and intradermal test) and oral provocation test as appropriate.
  Arms: Detailed penicillin allergy evaluation during pre-operative care

SUMMARY:
Use of first-line pre-operative antibiotic prophylaxis is the most effective measure to optimize perioperative outcomes. However, this is often not achieved due to unsubstantiated penicillin allergy labels. Penicillin allergy evaluation, when incorporated into routine pre-operative assessment, is potentially effective in optimizing choice of surgical prophylaxis. Despite the encouraging data mentioned above, there is a lack of randomized trials or local data to support this practice.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* planned for clean or clean-contaminated elective surgeries
* labelled allergy to penicillin group antibiotics on electronic patient record (ePR)

Exclusion Criteria:

* multiple antibiotic allergy
* history of severe cutaneous adverse reactions or other severe non-IgE-mediated hypersensitivity (e.g. haemolytic anaemia, organ dysfunction, serum sickness) due to beta-lactam antibiotics
* on systemic immunosuppressants
* pregnancy
* active or uncontrolled chronic urticaria
* mentally incompetent for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Use of first-line antibiotic | from the date of randomization up to 3 months
  The primary endpoint is use of first-line antibiotic for surgical prophylaxis according to local guideline .

SECONDARY OUTCOMES:
Antibiotic related adverse events | from the date of randomization up to 3 months
  Antibiotic related adverse events include: 1) any new symptoms reported by patients, or 2) abnormalities in blood tests that are compatible with known side effects of antibiotics given and that occurred after initiation of antibiotics.
Surgical site infection | from the date of randomization up to 30 days
  SSI is defined as an infection that occurs within 30 days after surgery in the part of the body where the surgery took place.
Colonization of multi-drug resistant organisms | from the date of randomization up to 3 months
  Multi-drug resistant organisms include methicillin resistant Staphylococcus aureus (MRSA), extended spectrum beta-lactamase (ESBL) producing Enterobacterales, carbapenem resistant Enterobacterales (CRE), multi-drug resistant Acinetobacter species (MDRA), multi-drug resistant Pseudomonas aeruginosa (MRPA), and vancomycin resistant Enterococci (VRE).
Length of stay | from the date of hospital admission up to hospital discharge or one year whichever earlier
  Length of hospital stay in this episode
All-cause mortality during hospital stay | form the date of randomization up to hospital discharge and from the date of randomization up to 3 months
  All-cause mortality during hospital stay and within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong